CLINICAL TRIAL: NCT05889650
Title: External Lumbar Drainage to Abort Severe Traumatic IntraCranial Hypertension: A Phase 1 Randomized, Allocation-concealed, Open-label, Safety and Feasibility Clinical Trial
Brief Title: External Lumbar Drainage to Reduce ICP in Severe TBI: a Phase 1 Clinical Trial
Acronym: ELASTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brain Trauma Foundation (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); University of Kansas (Other); The Cleveland Clinic (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Halinder Mangat, Director of Research, Brain Trauma Foundation
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 23-17380
Record Dates: First submitted 2023-05-20; First posted 2023-06-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Severe Traumatic Brain Injury; Intracranial Hypertension
Keywords: Traumatic brain injury; intracranial pressure; intracranial hypertension; lumbar drainage
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension

STUDY DESIGN:
Intervention Model Description: 2-stage randomization
Who Masked: Outcomes Assessor
Masking Description: Unaware of randomisation arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1st stage - prophylactic (Experimental): External lumbar drainage @15mmHg if intracranial pressure is not raised on admission
  Interventions: Procedure: External Lumbar drainage
- 2nd stage - treatment (Experimental): External lumbar drainage @20mmHg if / when intracranial pressure >20mmHg and tier 1 therapies cannot achieve ICP<20mmHg
  Interventions: Procedure: External Lumbar drainage
- Usual treatment (No Intervention): Usual treatment as per SIBICC algorithm

INTERVENTIONS:
Procedure: External Lumbar drainage — ELD @ 15 or 20mmHg based on intervention arm with maximum of 10ml/hour drainage
  Arms: 1st stage - prophylactic; 2nd stage - treatment

SUMMARY:
The goal of this phase 1 randomized controlled safety and feasibility clinical trial are to determine the safety of external lumbar drainage (ELD) in select patients with severe Traumatic Brain Injury (TBI). The main questions it aims to answer are (i) if ELD is feasible and (ii) safe to perform in severe TBI patients who have radiological evidence of patent basal cisterns and midline shift <5mm without increasing the risk of neurological worsening or cerebral herniation.

All participants will receive routine usual care. The study group will additionally have ELD for cerebrospinal fluid (CSF) drainage. A comparison will be made between the usual treatment plus ELD (interventional) groups, and the usual treatment (control) groups on incidence rate of neurological worsening or cerebral herniation events, and whether total hours with raised intracranial pressure (ICP) are different.

DETAILED DESCRIPTION:
This is a randomized controlled trial to determine the safety and feasibility of external lumbar drainage (ELD) of cerebrospinal fluid (CSF) as an adjunct to existing treatments to lower brain pressure, in select patients suffering severe traumatic brain injury (TBI). This trial is funded by the Department of Defense, Uniformed Services University of Health Sciences, Center for Neuroscience and Regenerative Medicine (CNRM).

Following a severe TBI, the brain swells and the pressure in the cranium rises causing further brain injury, The goal of treatment of such patients is to use treatments that lower brain swelling or pressure - directly by removing blood clots or indirectly by trying to lower the volume of contents in the cranium, viz. CSF or blood. Routinely a drain is placed in the skull to drain CSF out to provide space for brain swelling, thus keeping intracranial pressure (ICP) low. In some instances, all treatments available are unable to control swelling and the skull may need to be removed from one side, and in spite of this patients may die or suffer severe neurological injury and remain disabled.

Several non-randomized studies have shown that ELD is very effective in lowering intracranial pressure (ICP) in an immediate and lasting manner. While historical concerns remain that the brain may shift downwards causing herniation, this is not supported by recent studies. However, due to the historic nature of such teachings, some physicians may not use this potentially effective treatment in treating severe TBI patients with high ICP.

Therefore, in this trial we will determine the safety ELD in treating severe TBI patients, in a randomized controlled manner, whereby two-thirds of the patients will be randomized to routine usual treatments and either early or late ELD, and a third to only routine usual treatments. The patient randomized to ELD will receive this in addition to all other usual treatments, and no available treatment will be withheld

The secondary objectives are to determine if routine quantitative pupillometry can be used for safety determination and monitoring of ELD by evaluating:

1. Correlation with ELD safety score
2. Temporally changes prior to occurrence of any 'critical neuro-worsening events

Comparison / Usual treatment All participants will undergo usual treatment as per evidence- and guidelines-based Seattle International Severe Traumatic Brain Injury Consensus Conference (SIBICC) algorithm (36, 71). Routine non-invasive automated infra-red pupillometry will be performed bilaterally every hour as part of routine neurological checks for neuro-worsening in addition to hourly Glasgow Coma Scale (GCS) score checks and other routine intensive care unit (ICU) protocols. No treatment will be withheld. ICP monitoring will be performed with intra-parenchymal monitor or external ventricular drainage (EVD) as per local protocols.

RISKS TO HUMAN SUBJECTS:

The assessments for this study involve risk and benefits to patients in excess of routine standard of care treatment. The risks related to the intervention i.e. placement of lumbar drain and drainage of CSF, are critical neurological worsening events related to cerebral herniation such as decrease in GCS score, development of new motor deficit, or rarely death. These events will be recorded for all patients and prompt treatment will be instituted accordingly, including an emergent computed tomography (CT) scan (36). Clinical protocols exist at all neurotrauma ICUs for such neuro-worsening events and neurointensivists and neurotrauma surgeons are well placed to manage them medically or surgically in routine care of severe TBI patients.

Background 'Event rate' for critical neuro-worsening events with usual treatment: To estimate background 'event rate' of critical neuro-worsening events, we analyzed the Brain Trauma Foundation (BTF)-New York State TBI-trac® registry from 1997-2004, with 4789 TBI patients, of which 3590 had CT data and 2616 were between the age of 18-65 years. When inclusion / exclusion criteria for age and CT findings were applied, 50.3% of these were eligible for the study. The mean incident risk of having new pupillary asymmetry at any point after admission was 22.0% (95% confidence intervals (CI): 19.9-24.3%), risk of motor worsening was 18.0% (95% CI: 12.6-25.0%) for those with motor score 1-4, and 16.4% (95% CI: 12.1-21.9%) for all motor scores with deterioration. Finally, risk of 2-week mortality was 22.4% (95% CI 20.2-24.8%). This data provides us with an expected event rate, though the comparison will still be made between control and intervention arms of the study, per protocol. Given the high incidence of these events occurring as natural history of the disease, they will be classified as anticipated Serious adverse events (SAEs).

Human Subjects Protections:

Pressure and Volume protected lumbar CSF drainage: In the studies reviewed, ELD was set to drain at 0-20 mmHg or drained at fixed volume. In order to increase safety, we will perform ELD in patients without high ICP at 15 mmHg and those with high ICP at 20 mmHg and additionally volume-limit drainage to 10 ml/hour.

Procedure safety:

Indication:

ELD will be utilized as the first intervention in the 2nd tier of SIBICC protocol, which will invariably be preceded by gradual increase in ICP. As per SIBICC protocol, a CT scan will be obtained prior to advancement to 2nd tier and ELD placement.

Contra-indications:

ELD will NOT be utilized to lower ICP during sudden ICP crises associated with neuro-worsening. Hypertonic saline, mannitol, hyperventilation, and review for surgery will be utilized as per clinical routine.

ELD will NOT be placed in lieu of an EVD. ELD will NOT be performed in patients undergoing hemicraniectomy.

Safety Monitoring: Given the greatest risk of neuro-worsening from herniation is soon after drainage is commenced, all patients will undergo automated pupillometry for pupillary size, symmetry, light reactivity and neurological pupillary index (NPI) every 15 minutes for 1 hour following ELD placement and start of CSF drainage. Following the first hour, pupillometry will be performed hourly. If NPI drops by 1 point within the 1st hour, a head CT may be obtained to review any craniocaudal shift.

SAFETY REPORTING: All unanticipated SAEs will be reported to the steering committee, local site institutional research boards (IRBs) as well as the overall IRB, within 24 hours. Anticipated SAE and adverse events (AEs) will be reported in annual reports.

Data Safety and Monitoring Board (DSMB):

A DSMB of a pool of 7 experienced trauma neurosurgeons and neurointensivists of international standing, will review every neuro-worsening events, as defined above, in each arm of the study. The DSMB will meet every 6 months to review anticipated SAEs. DSMB will review unanticipated SAE including deaths within 48 hours, and will make determinations of association of unanticipated adverse events with interventions.

Potential benefits of the proposed research to participants:

As this is an interventional study, the research participants may gain direct benefit or suffer harm. At conclusion of the study, the overall results will be included in a summary report mailed to all participants. In the field of TBI management, this study has potential benefits in treating post-traumatic intracranial hypertension, which is the main mechanism of neurological deterioration following severe TBI and improving functional outcome for participants.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years age
2. Glasgow Coma Scale (GCS) 3-8
3. Pupils symmetric and bilaterally reactive
4. Midline shift ≤5mm at the level of foramen of Monro on admission or post-operative brain CT
5. Patent (complete or partial) quadrigeminal cisterns on admission or post-operative brain CT
6. First randomization and intervention may be commenced within 24 hours of injury
7. ELD safety score ≥5

Exclusion Criteria:

1. GCS >8
2. Cisterns on CT completely effaced
3. Midline shift on CT >5mm
4. GCS 3 with dilated and fixed pupils
5. Uncal or tonsillar herniation on admission or post-operative brain CT
6. Temporal lobe contusions
7. Penetrating TBI
8. Primary hemicraniectomy
9. Pregnancy
10. Prisoners
11. Patients previously lacking capacity to consent or refuse treatment, or with advanced directives to forego aggressive care
12. Pre-existing conditions affecting functional status or life expectancy to less than 1 year
13. Contra-indications for ELD placement: coagulopathy, use of anticoagulants or anti-thrombotics, thrombocytopenia <50,000, or severe spinal deformity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of ELD in selected Severe TBI patients | 10 days
  Rate of occurrence of herniation events or death in 3 arms
Feasibility of ELD in selected Severe TBI patients | 10 days
  Proportion of patients able to undergo treatment as per randomised arm

SECONDARY OUTCOMES:
Reduction in ICP burden using ELD in selected severe TBI patients | 10 days
  Total number of hours with ICP>20mmHg
Utility of automated pupillometry to predict safety of ELD | 10 days
  worsening of Pupillometry based reactivity index in 6 hours preceding herniation events with occurrence of such events

CONTACTS AND LOCATIONS:
Overall Officials: Halinder S Mangat, MD MSc, Principal Investigator — Brain Trauma Foundation; Kansas University Medical Center Research Institute; Jamshid Ghajar, MD PhD, Principal Investigator — Brain Trauma Foundation; Gregory Hawryluk, MD PhD, Principal Investigator — Cleveland Clinic Foundation, Brain Trauma Foundation; Bradley Dengler, MD, Study Chair — Military Traumatic Brain Injury Initiative, Uniformed Services University
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Badhiwala J, Lumba-Brown A, Hawryluk GWJ, Ghajar J. External Lumbar Drainage following Traumatic Intracranial Hypertension: A Systematic Review and Meta-Analysis. Neurosurgery. 2021 Aug 16;89(3):395-405. doi: 10.1093/neuros/nyab181. PMID 34171100
- [Background] Ginalis EE, Fernandez LL, Avila JP, Aristizabal S, Rubiano AM. A review of external lumbar drainage for the management of intracranial hypertension in traumatic brain injury. Neurochirurgie. 2022 Feb;68(2):206-211. doi: 10.1016/j.neuchi.2021.05.004. Epub 2021 May 26. PMID 34051245
- [Background] Bauer M, Sohm F, Thome C, Ortler M. Refractory intracranial hypertension in traumatic brain injury: Proposal for a novel score to assess the safety of lumbar cerebrospinal fluid drainage. Surg Neurol Int. 2017 Nov 1;8:265. doi: 10.4103/sni.sni_98_17. eCollection 2017. PMID 29184716
- [Background] Llompart-Pou JA, Abadal JM, Perez-Barcena J, Molina M, Brell M, Ibanez J, Raurich JM, Ibanez J, Homar J. Long-term follow-up of patients with post-traumatic refractory high intracranial pressure treated with lumbar drainage. Anaesth Intensive Care. 2011 Jan;39(1):79-83. doi: 10.1177/0310057X1103900113. PMID 21375095
- [Background] Murad A, Ghostine S, Colohan AR. A case for further investigating the use of controlled lumbar cerebrospinal fluid drainage for the control of intracranial pressure. World Neurosurg. 2012 Jan;77(1):160-5. doi: 10.1016/j.wneu.2011.06.018. Epub 2011 Nov 15. PMID 22154151
- [Background] Abadal-Centellas JM, Llompart-Pou JA, Homar-Ramirez J, Perez-Barcena J, Rossello-Ferrer A, Ibanez-Juve J. Neurologic outcome of posttraumatic refractory intracranial hypertension treated with external lumbar drainage. J Trauma. 2007 Feb;62(2):282-6; discussion 286. doi: 10.1097/01.ta.0000199422.01949.78. PMID 17297313
- [Background] Tuettenberg J, Czabanka M, Horn P, Woitzik J, Barth M, Thome C, Vajkoczy P, Schmiedek P, Muench E. Clinical evaluation of the safety and efficacy of lumbar cerebrospinal fluid drainage for the treatment of refractory increased intracranial pressure. J Neurosurg. 2009 Jun;110(6):1200-8. doi: 10.3171/2008.10.JNS08293. PMID 19249925
- [Background] Hawryluk GWJ, Aguilera S, Buki A, Bulger E, Citerio G, Cooper DJ, Arrastia RD, Diringer M, Figaji A, Gao G, Geocadin R, Ghajar J, Harris O, Hoffer A, Hutchinson P, Joseph M, Kitagawa R, Manley G, Mayer S, Menon DK, Meyfroidt G, Michael DB, Oddo M, Okonkwo D, Patel M, Robertson C, Rosenfeld JV, Rubiano AM, Sahuquillo J, Servadei F, Shutter L, Stein D, Stocchetti N, Taccone FS, Timmons S, Tsai E, Ullman JS, Vespa P, Videtta W, Wright DW, Zammit C, Chesnut RM. A management algorithm for patients with intracranial pressure monitoring: the Seattle International Severe Traumatic Brain Injury Consensus Conference (SIBICC). Intensive Care Med. 2019 Dec;45(12):1783-1794. doi: 10.1007/s00134-019-05805-9. Epub 2019 Oct 28. PMID 31659383